CLINICAL TRIAL: NCT01264315
Title: Safety And Efficacy Of Lenalidomide As Maintenance Therapy In Patients With Newly Diagnosed Multiple Myeloma Following A Tandem Autologous-Allogeneic Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-MM-GITMO-413; 2008-004529-41 (EudraCT Number)
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Multiple Myeloma
Keywords: Lenalidomide; Tandem Autologous-Allogeneic Transplant
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide in maintenance (Other)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide will be started at 6 months post-allotransplant at 10 mg/day continuously in all patients:
  * absolute neutrophil count >1x109/L without growth factors
  * platelet count >75x109/L without transfusion support
  * calculated/measured creatinine clearance: ≥20mL/minute
  * total bilirubin <2 x the upper limit of normal
  * AST (SGOT) and ALT (SGPT) <2.5 x upper limit of normal
  * <1mg/kg/day of prednisone, and no more than 2 immunosuppressive drugs other than steroid to control GVHD
  Treatment will be continued without interruption, unless not tolerated, until unacceptable adverse events or progressive disease occur. In case of disease progression occurring before the start of lenalidomide, the patient will be withdrawn from study and treated according to the center preference. Lenalidomide will be discontinued in patients achieving and maintaining molecular remission for 2 consecutive controls at least 6 weeks apart.

SUMMARY:
Rationale: We recently reported a study where overall and event free survivals in newly diagnosed myeloma patients receiving an autologous transplant followed by an allograft from an HLA-identical sibling were superior as compared to those undergoing a double autologous transplant. A larger multicenter study by the Gruppo Italiano Trapianti di Midollo (GITMO), co-ordinated by our group and recently closed, employing a tandem auto-allo approach in newly diagnosed patients confirmed the achievement of prolonged event free and overall survival. Importantly, the achievement of at least very good partial remission at the time of allografting conferred a significant advantage in both event-free-survival (HR 0,23, CI 0,11-0,48; p=0,0001) and overall survival (HR 0,26; CI 0,09-0,79; p=0,02). Moreover, recent advances in the understanding of the pathogenesis of multiple myeloma have identified specific signalling pathways that have become targets for biologically-based drugs such as thalidomide, bortezomib and lenalidomide and employed in several trials, including after allograft. The aim of the current proposal is to combine the post-transplant efficacy of graft-vs.-myeloma with the anti-myeloma effect of lenalidomide in newly diagnosed myeloma patients with an HLA-identical sibling treated with a tandem autograft-allograft approach. Maintenance/consolidation of the response may be a key factor to further improve rate of clinical and molecular (as a prelude to cure) remissions and prolong overall and event free survivals after allografting. We would like to investigate the safety and efficacy of lenalidomide as consolidation/maintenance therapy in patient undergoing tandem autologous-allogeneic transplant.

Objectives of study: To evaluate 1) toxicity and tolerability of lenalidomide after allografting; 2)To evaluate efficacy of lenalidomide in inducing complete remission, defined as negative immunofixation, 12 months after allografting; 3) overall-survival; 4) event-free survival; 5) molecular remission rate. Furthermore we plan to compare molecular remission rate in patients treated with lenalidomide after tandem auto-allo transplant and after double autologous transplant and to monitor minimal residual disease in patients achieving clinical CR with lenalidomide.

Patient Selection: Patients with newly diagnosed multiple myeloma with an HLA identical sibling suitable for PBSC donation will be included. Complete cytogenetic analysis at diagnosis will be required. The patient must have the capacity to give informed consent. Age >18 and < 65. Negative pregnancy test and willing to use contraceptive techniques during and for 12 months following treatment is required. Only very unfitted patients will be excluded.

Treatment plan: Lenalidomide will be started at 6 months post-allotransplant at the dose of 10 mg/day continuously in all patients (unless in molecular CR), if the following conditions are present:

* absolute neutrophil count > 1 x 109/L without the use of growth factors;
* platelet count > 75 x 109/L without transfusion support;
* calculated or measured creatinine clearance: ≥ 20 mL/minute;
* total bilirubin < 2 x the upper limit of normal,
* AST and ALT < 2.5 x upper limit of normal
* less than 1 mg/kg/day of prednisone, and no more than 2 immunosuppressive drugs other than steroid to control GVHD (if more immunosuppression is required to control GVHD, the maintenance therapy with lenalidomide will be held until this criteria will be satisfied) Treatment will be continued without interruption, unless not tolerated, until unacceptable adverse events are experienced or progressive disease occurs. Moreover, lenalidomide will be discontinued in patients who achieve and maintain molecular remission for 2 consecutive controls at least 6 weeks apart.

Safety section - dose modification plan: During the study patients will be monitored for the occurrence of side effects. Toxicity events will be graded according to the NCI toxicity criteria. In case of severe toxicity, the lenalidomide dose will be reduced or withheld as outlined in the protocols.

Statistical section: - Total patient sample size: 53. This is a phase 2 study designed according to a Simon's two-stage Minimax Design. An early stopping rule will be established to interrupt the study in case of futility (a non satisfactory response rate). In stage I 27 patients will be enrolled; if < 14 complete remissions will be observed, the trial will be stopped. In stage II 26 more patients will be enrolled. If ≥ 32 responses will be observed, it will be concluded that the lenalidomide maintenance is active in increasing the complete remission rate after auto-allograft.

Analysis plan: Toxicity monitoring will be incorporated into the study design by requiring that the trial be terminated after an initial stage if the number of observed toxicities (treatment related deaths) is excessive.

DETAILED DESCRIPTION:
A. Pre-transplant phase: Induction Therapy

Patients will start induction treatment with lenalidomide and dexamethasone (RD) for 4 cycles every 28 days (as was detailed also in the GIMEMA protocol RV-MM-PI-209):

* Lenalidomide will be given orally at the dose of 25 mg/day for 21 days followed by a 7 day rest period (day 22 to 28),
* Dexamethasone will be given orally at the dose of 40 mg on days 1, 8, 15 and 22 every 28 days.

If a patient relapses during RD before the end of the 4th cycle, the induction treatment may be held and stem cell collection may be attempted with cyclophosphamide according to physician willing.

For dose reduction during induction therapy see Appendix O. Antithrombotic prophylaxis as per protocol RV-MM-PI-209. For patients not previously enrolled in protocol RV-MM-PI-209, we recommend prophylaxes with aspirin for patients without additional thrombotic risk factors, and low molecular weight heparin (LMWH) 100 U/kg for the others.

Otherwise, induction schemas are accepted provided thalidomide, lenalidomide or bortezomib, alone or in combination, are included.

B. Peripheral Blood Stem Cell (PBSC) Mobilization and collection

After 1-2 months from the completion of the last induction course, patients will undergo PBSC mobilization with cyclophosphamide 4 g/m2 and G-CSF (10 ug/kg/day starting at day 5 until completion of PBSC collection) to collect an adequate number of PBSC (4 to 10 x 106/kg CD 34+ cells). Patients who fail to collect the minimum of 4 x 106/kg CD 34+ cells will receive a second course of cyclophosphamide for a second mobilization attempt. Patients who fails to collect a minimum of 4 x 106/kg CD 34+ will be withdrawn from the study.

C. High-Dose Melphalan / Autologous PBSC Transplant

High dose melphalan will be given 4 to 8 weeks after high dose cyclophosphamide.

1. Melphalan will be administered at a cumulative dose of 200 mg/m2. This will be given in one dose infused on day -2. Dose will be calculated according to the participating institutional standard practice for using body weight. High dose Melphalan is administered via a central catheter as per single center procedure.
2. Peripheral Blood Stem Cell or Bone Marrow Infusion: Infuse > 2 x 106 CD 34+ cells /kg, hydration requirements, and pre-medication per guidelines of the institution.
3. G-CSF: Administer G-CSF 5 ug/kg/day subcutaneously or intravenously from day +3 until ANC >1000 for 3 days.

D. Allogeneic transplant phase: Non-myeloablative PBSC Allografting

Pre-conditioning Upon recovery from high-dose melphalan, between 40-120 days post autografting (preferably within 60 days) patients will proceed to nonmyeloablative allograft. If indicated, radiation to high risk skeletal lesions may be given pre-transplant. If interval exceeds 120 days, present to PCC for discussion and approval.

Recovery from high-dose melphalan will be defined by patients achieving the following clinical criteria after receiving high dose melphalan:

1. mucositis and gastrointestinal symptoms resolved, off hyperalimentation and intravenous hydration;
2. have completed steroids for autologous GVHD;
3. LFT / renal function values within the inclusion criteria for initial autograft;
4. off IV antibiotics and amphotericin for documented infections;
5. patients should be CMV antigenemia negative;
6. if patients have experienced CMV infection post-autograft, they must have completed therapy with Ganciclovir or Foscarnet and have been off this therapy for > two weeks and remain CMV antigenemia negative;
7. should have completed administration of any radiotherapy;
8. any patient who does not fulfill these criteria, can be discussed with the principle investigator for recommendations as to the timing of the allograft.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed multiple myeloma patients with an HLA identical sibling suitable for PBSC donation and treated in induction with thalidomide or bortezomib or lenalidomide conteining regimes.
2. Complete cytogenetic analysis at diagnosis, including FISH analysis for chromosome deletions 13 and 17, and translocations (4;14) (11;14) and (14;16).
3. The patient must have the capacity to give informed consent.
4. Age >18 and < 65
5. If female, the patient is either postmenopausal since at least 24 consecutive months or surgically sterilized or she agrees to practice sexual abstinence or to use two reliable methods for contraception (e.g. a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide) for the duration of study
6. If male, the patient agrees to practice sexual abstinence or to use a latex condom during any sexual contact with women of childbearing potential for the duration of study
7. Negative pregnancy test

Exclusion Criteria:

1. Karnofsky score less than 60 (see appendix C), unless due solely to myeloma
2. Left ventricular ejection fraction less than 40%, or symptomatic coronary artery disease or other cardiac failure requiring therapy
3. Bilirubin greater than 2 X the upper limit of normal, or SGPT and SGOT > 4 X the upper limit of normal
4. DLCO < 40% (corrected) or receiving continuous supplemental oxygen.
5. Creatinine clearance < 40 cc/min at the time of initial autografting evaluation.
6. Patients with poorly controlled hypertension
7. Patients with active non-hematologic malignancies (except non-melanoma skin cancers).
8. Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a >20% risk of disease recurrence
9. Seropositive for HIV
10. Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment.
11. To evaluate toxicity and tolerability of lenalidomide after allografting
12. To evaluate efficacy of lenalidomide in inducing complete remission 12 months after allografting

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Lenalidomide toxicity and tolerability after allografting | 6 years
  To evaluate toxicity and tolerability of lenalidomide after allografting.
Lenalidomide efficacy | 1 years
  To evaluate efficacy of lenalidomide in inducing complete remission, defined as negative immunofixation, 12 months after allografting.

SECONDARY OUTCOMES:
Overall survival | 6 years
Progression free survival | 6 years
Event free survival | 6 years
Molecular remission rate | 6 years
  To evaluate molecular remission rate, and to compare molecular remission rate in patients treated with lenalidomide after tandem auto-allo transplant and after double autologous transplant (study protocol RV-MM-PI-209): molecular remission is defined as the disappearance of the disease- and patient-specific molecular marker by polymerase chain reaction (PCR)-based assay, in both bone marrow and blood on two consecutive tests at least six weeks apart.
Minimal residual disease | 6 years
  To monitor minimal residual disease in patients achieving clinical CR with lenalidomide.

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Giaccone, MD, Principal Investigator — Division of Hematology - University of Torino - A.O.U. Città della Salute e della Scienza di Torino - Torino - Italy
Locations (1):
- A.O.U. Città della Salute e della Scienza di Torino, Torino, Italy